CLINICAL TRIAL: NCT04333264
Title: Clinical Analysis of Suction Drainage in Cementless Hip Replacement - a Prospective Randomized Study
Brief Title: Clinical Analysis of Suction Drainage in Cementless Hip Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bartosz Paweł (Other)
Responsible Party: Sponsor-Investigator, Bartosz Paweł, Principal investigator, Prof A Gruca Teaching Hospital
Organization: Prof A Gruca Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1/032016
Record Dates: First submitted 2020-03-30; First posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Arthropathy of Hip
Keywords: hip; arthroplasty; suction; drainage
MeSH Terms: interventions — Suction

STUDY DESIGN:
Intervention Model Description: Two groups of patients with or without closed suction drainage after primary total hip arthroplasty.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- suction drainage (Active Comparator): Patients will be dived with randomization in to two groups: with and without closed suction drainage after primary total hip arthroplasty
  Interventions: Procedure: suction drainage
- no suction drainage (Active Comparator): Patients will be dived with randomization in to two groups: with and without closed suction drainage after primary total hip arthroplasty
  Interventions: Procedure: no suction drainage

INTERVENTIONS:
Procedure: suction drainage — After primary total hip arthroplasty closed suction drainage will be used.
  Arms: suction drainage
Procedure: no suction drainage — After primary total hip arthroplasty closed suction drainage won't be used.
  Arms: no suction drainage

SUMMARY:
Randomized prospective study assessing suction drainage in total hip arthroplasty. Group without drainage, 50 hips, compared with group with suction drainage, 50 hips. Both groups will be asses clinically (ROM scale, VAS), laboratory and radiology (USG). In the actually literature there are no benefits using closed suction drainage after primary total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* age between 30-80
* primary hip osteoarthritis

Exclusion Criteria:

* secondary hip osteoarthritis
* autoimmune disease
* congenital or secondary coagulopathy
* vein or artery thrombosis
* renal or liver failure
* cemented or hybrid alloplasty,
* no consent from the patient

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Hip hematoma size in USG | 3 days after surgery
  Size in millimeters fluid collection in supine position above femoral neck.
Hemoglobin levels | 3 days after surgery
  Hb levels after surgery, difference between two groups
C-reactive protein levels | 3 days after surgery
  C-reactive protein levels after surgery, difference between two groups
Visual Analog Scale punctation | 3 day after surgery
  Pain level after surgery in Visual Analog Scale scale 0-10 pts. where 0-no pain, 10-most painful.
Hip range of movement | 3 days after surgery
  Differences between hip ROM after surgery
Wound exudation | 3 days after surgery
  Assessing wound dehiscence after surgery, 1-exudation appear, 0-dry dressing
Soft tissue hematoma | 3 days after surgery
  USG hematoma appearance in soft tissue around the hip
Intraoperative bleeding | 1 day
  All amount of blood loss intraoperative with hidden bleeding, with use of Gross formula.
Blood transfusion | 14 days after surgery
  Need of blood transfusion after operation

SECONDARY OUTCOMES:
Infection | 30 days after surgery
  Superficial or deep infection after surgery
Deep vein thrombosis | 30 days after surgery
  Occurrence lower limb thrombosis after surgery
Readmission | 30 days after surgery
  Need to readmission after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Pawel Bartosz, Principal Investigator — Prof. A. Gruca Teaching Hospital in Otwock

REFERENCES:
- [Derived] Bartosz P, Marczynski W, Para M, Kogut M, Bialecki J. Comparative study of suction drainage placement in cementless hip replacement among patients undergoing extended thromboprophylaxis: a prospective randomized study. BMC Musculoskelet Disord. 2021 Aug 13;22(1):688. doi: 10.1186/s12891-021-04583-0. PMID 34389016